CLINICAL TRIAL: NCT05561114
Title: Paclitaxel Coated Balloon for the Treatment of Chronic bEnigN sTricture- Esophagus
Acronym: PATENT-E
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GIE Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR2052
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Stricture
Keywords: esophageal stricture; drug coated balloon; DCB; paclitaxel coated balloon
MeSH Terms: conditions — Esophageal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- GIE Medical ProTractX3 TTS DCB (Experimental): The ProTractX3 Drug-coated balloon is a 0.035" guidewire compatible over-the-wire catheter.
  Interventions: Combination Product: GIE Medical ProTractX3 TTS DCB
- Control (Active Comparator): Standard of Care Endoscopic Dilation
  Interventions: Other: Control

INTERVENTIONS:
Combination Product: GIE Medical ProTractX3 TTS DCB — Paclitaxel Coated Balloon
  Arms: GIE Medical ProTractX3 TTS DCB
Other: Control — Standard Endoscopic Dilation
  Arms: Control

SUMMARY:
To evaluate the safety and efficacy of the ProTractX3™ DCB for the treatment of benign esophageal strictures.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22 years
2. Diagnosis of a benign esophageal stricture with at least 2 previous dilations
3. Ogilvie Dysphagia Score of ≥2
4. Minimum esophageal lumen diameter <13 mm
5. Willing and able to complete protocol required follow-up visits
6. Willing and able to provide written informed consent
7. Strictures ≤5cm in total length
8. Target benign esophageal stricture etiologies include:

   1. Peptic stricture,
   2. Schatzki's ring,
   3. Stricture due to prior infection,
   4. Post-procedural (e.g. ESD/EMR/RFA/Cryo) stricture
   5. Post surgical (e.g. anastomotic), including post curative esophagectomy with or without prior neoadjuvant chemoradiation therapy

Exclusion Criteria:

1. Two or more clinically significant (e.g. non-traversable) strictures with total length >5cm or unable to be treated with a single balloon.
2. Female subjects who are pregnant or breastfeeding or plan to become pregnant in next 12 months
3. Contraindication to endoscopy, anesthesia or deep sedation
4. Benign esophageal stricture due to extrinsic esophageal compression, caustic ingestion, lichen planus, and purely radiation induced strictures post head/neck cancer treatment.
5. History of diagnosis of eosinophilic esophagitis (EoE)
6. Signs or suspicion of a malignant esophageal stricture NOTE: If stricture is suspicious for malignancy based on clinical or endoscopic presentation, malignancy must be excluded by biopsy prior to enrollment. Subjects with a history of invasive esophageal cancer should have recurrence excluded by advanced imaging (e.g. CT/PET scan) and biopsy within 6 months of enrollment.
7. Diagnosis of metastatic cancer of any type that is not considered in remission or non-metastatic cancer that may require radiation treatment in the neck or thoracic region NOTE: A prior diagnosis of esophageal cancer is acceptable if considered in remission and recurrence has been excluded by advanced imaging and biopsy within 6 months of enrollment.
8. Suspected perforation of gastrointestinal tract
9. Inability to pass guidewire across stricture
10. Active systemic infection
11. Allergy to paclitaxel or structurally related compounds
12. Severe coagulation disorders or current use of anticoagulant or antiplatelet medication that cannot be safely managed per recommended guidelines prior to the index procedure
13. Chronic systemic steroid use for any medical conditions unless subject is willing to undergo a 4-week washout and discontinue steroid use
14. Received steroid injections into target stricture in the last 8 weeks.
15. Stricture not amenable to endoscopic dilation to ≥ 18 mm in the opinion of the investigator
16. Current use of nasal or oral feeding tube unless tube is removed prior to baseline assessments and subject maintains normal swallowing function.
17. Acute stricture condition that requires emergent procedure (e.g. immediate dilation)
18. Stricture complicated with abscess, fistula, deep ulceration, perforation, leakage or varices, or thrombosis, etc
19. Life expectancy of less than 24 months
20. Concurrent medical condition that would affect the investigator's ability to evaluate the patient's condition or could compromise patient safety, such as recent myocardial infarction, severe pulmonary disease, bleeding diathesis, large thoracic aneurysm, pharyngeal or cervical deformity, ongoing infection, etc
21. Current participation in another pre-market drug or medical device clinical study that has not reached it's primary endpoint.
22. Dysphagia related to primary motility disorders, such as achalasia, diffused esophageal spasm, ineffective esophageal motility (IEM), hypertensive lower esophageal sphincter, esophageal outlet obstruction, etc.
23. Active erosive esophagitis with a Los Angeles classification of Grade B-D at the time of endoscopy.
24. Significant esophageal dilation proximal to the stricture that, in the Investigator's opinion, may impact long-term esophageal motility.
25. Intolerant to effective acid suppression medication (e.g. proton pump inhibitors, H2 receptor antagonists)
26. Concurrent gastric and/or duodenal obstruction

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Treatment Success | 6 Months Post-Procedure
  1. The primary efficacy endpoint is freedom from stricture recurrence, measured as the time from Index procedure until stricture recurrence through 6 months post-procedure. Stricture recurrence is defined as an esophageal diameter <13mm as measured using a functional luminal imaging probe, or clinically driven reintervention at the treated area within 6 months post-procedure as determined by the Clinical Events Committee
Primary Safety Outcome | 30 Days Post-Treatment
  Incidence of device- and/or procedure-related Major Adverse Events (MAEs) (Death, perforation of the esophagus, bleeding requiring intervention or transfusion)

SECONDARY OUTCOMES:
Annualized Rate of Reintervention | Annually
  The annualized reintervention rate is defined as the annualized number of clinically driven interventions and will be assessed by comparing the annualized rate per patient year between groups using a test of Poisson rates.
Diameter Improvement at 6 months | 6 Months Post-Procedure
  The minimum esophageal stricture diameter will be assessed by a functional luminal imaging probe (EndoFLIP) during endoscopy and compared between the Test and Control arms. The minimum esophageal stricture diameter will be measured at baseline and during the 6-month follow-up, or at the time of a reintervention if one occurs prior to 6 months.
Clinical Responder Rate at 6 months | 6 Months Post-Procedure
Freedom from clinically driven target stricture reintervention through 6 months post-procedure | 6 Months Post-Procedure
Freedom from symptom recurrence through 6 months post-procedure | 6 Months Post-Procedure

OTHER OUTCOMES:
Secondary Patency | Time between the index procedure to the second clinically driven intervention
Technical Success | Procedure
Annualized rate of dilations before and after treatment | Annually
Improvement in time between dilations | Between Dilations
Improvement in Ogilvie Dysphagia Score at each follow-up | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Improvement in Dysphagia Handicap Index score at each follow-up | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Stricture characteristics per functional imaging | Between Dilations
Number of esophageal dilation procedures through each follow up | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Freedom from clinically driven reintervention through each follow-up | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Freedom from symptom recurrence through each follow-up | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
VAS for pain scores through 30-day follow-up | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years
Composite EQ-5D quality of life scores at each follow-up | 30 days, 3 months, 6 months, 12 months, and annually thereafter through 5 years

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Birmingham Gastroenterology Associates, Birmingham, Alabama
  - Honor Health, Scottsdale, Arizona
  - University of California, Irvine, Irvine, California
  - Gastro Care Institute, Lancaster, California
  - Cedars Sinai, Los Angeles, California
  - San Diego Gastroenterology, San Diego, California
  - University of Colorado Anschutz, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Borland-Groover, Jacksonville, Florida
  - Research Associates of South Florida, Miami, Florida
  - Hillcrest Medical Research, Orange City, Florida
  - Orlando Health, Orlando, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Rush University, Chicago, Illinois
  - Kansas Gastroenterology, LLC, Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Sierra Clinical Research, Las Vegas, Nevada
  - Rutgers University, Piscataway, New Jersey
  - New York Presbyterian Hospital- Columbia University Medical Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor St. Luke's Medical Center, Houston, Texas
  - TEN20 Clinical Research, Plano, Texas
  - The University of Utah, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No